CLINICAL TRIAL: NCT06121830
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group, Phase 3, Therapeutic Confirmatory Clinical Trial to Evaluate the Efficacy and Safety of DWP14012 in Patients With Non-erosive Gastroesophageal Reflux Disease
Brief Title: Study to Evaluate the Efficacy and Safety of DWP14012 in Patients With Non-Erosive Gastroesophageal Reflux Disease (NERD)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWP14012311
Record Dates: First submitted 2023-10-16; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Non-erosive Reflux Disease; Non-Erosive Gastro-Esophageal Reflux Disease; Non-Erosive Esophageal Reflux Disease
Keywords: NERD
MeSH Terms: conditions — Non-Erosive Reflux Disease | interventions — fexuprazan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DWP14012 20mg (Experimental): Once daily with water regardless of meals without chewing or crushing for 4 weeks.
  Interventions: Drug: DWP14012 20mg
- DWP14012 40mg (Experimental): Once daily with water regardless of meals without chewing or crushing for 4 weeks.
  Interventions: Drug: DWP14012 40mg
- Placebo (Placebo Comparator): Once daily with water regardless of meals without chewing or crushing for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DWP14012 20mg — DWP14012 20mg, tablet, orally, once daily for up to 4 weeks
  Arms: DWP14012 20mg
Drug: DWP14012 40mg — DWP14012 40mg, tablet, orally, once daily for up to 4 weeks
  Arms: DWP14012 40mg
Drug: Placebo — Placebo, tablet, orally, once daily for up to 4 weeks
  Arms: Placebo

SUMMARY:
This study is designed to determine the efficacy and safety of DWP14012 compared to a placebo following a once-daily oral dose of DWP14012 at 20 mg, 40 mg, or placebo for 4 weeks in patients with NERD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged 19 to 75 years, both inclusive, at the date of obtaining informed consent
2. Subjects with no mucosal break(s) according to Los-Angeles grade on EGD performed at the same site within 2 weeks prior to Visit 1
3. Subjects who have experienced heartburn for at least 12 weeks prior to Visit 1
4. Subjects who have completed all symptom assessments (heartburn, acid regurgitation) in the subject diary from 7 days to 1 day prior to Visit 2
5. Subjects who have experienced one of the following symptoms according to the symptom assessments in the subject diary from 7 days to 1 day prior to Visit 2
6. Subjects who have reported at least moderate burning sensation in the esophagus (behind the breastbone) for heartburn symptoms for at least 4 days
7. Subjects who have reported at least moderate pain in the esophagus (behind the breastbone) for heartburn symptoms for at least 4 days
8. Subjects who are capable of understanding the provided information and able to comply with all the study procedures including filling out the subject diary and questionnaire throughout the study
9. Subjects who voluntarily decide to participate in the study and sign the informed consent form

Exclusion Criteria:

1. Subjects who have Barrett's esophagus, gastroesophageal varix, viral/fungal gastrointestinal infection, esophagostenosis, ulcer stenosis, active peptic ulcer, gastrointestinal bleeding, or a malignant tumor identified on EGD performed within 2 weeks prior to Visit 1
2. Subjects who have warning symptoms of malignant gastrointestinal tract diseases such as odynophagia, severe dysphagia, bleeding, weight loss, anemia, or hematochezia at Visit 1 (However subjects who have additional warning symptoms besides typical symptoms of gastroesophageal reflux disease [GERD] may be included if the result of endoscopy, etc. is negative for the presence of tumor.)
3. Subjects with Zollinger-Ellison syndrome at Visit 1
4. Subjects with eosinophilic esophagitis at Visit 1
5. Subjects who are diagnosed with erosive GERD, acute upper gastrointestinal bleeding, gastric ulcer, or duodenal ulcer within 8 weeks prior to Visit 1
6. Subjects who are diagnosed with FD, FH, RH, primary esophageal motility disorder, IBS, and IBD within 12 weeks prior to Visit 1
7. Subjects who had a surgery to reduce gastric acid secretion, or gastric or esophageal surgery (e.g., gastrectomy, mucosal resection, etc.) (Except, simple perforation surgery and endoscopic resection of benign tumors)
8. Subjects who have a clinically significant disease of hepatic, renal, neurologic, respiratory, endocrine, hemato-oncologic, cardiovascular or urinary system at Visit 1
9. Subjects who have history of alcohol or other drug abuse within 1 year prior to Visit 1
10. Subjects diagnosed with malignant tumor within 5 years prior to Visit 1 (Subjects completely healed for ≥5 years from the last treatment without recurrence are allowed to be enrolled.)

    * Subjects with cured basal cell carcinoma of the skin or carcinoma in situ of the cervix are allowed to be enrolled regardless of time period
    * Subjects with a history of digestive malignant tumor are excluded regardless of the time period
11. Subjects who have or had bipolar disorder, anxiety disorder, panic disorder, somatoform disorder, personality disorder, or other clinically significant psychiatric disorders
12. Subjects with scleroderma (systemic sclerosis) or systemic lupus erythematosus
13. Subjects who have hypersensitivity, or medical history of clinically significant hypersensitivity, to any components of the IP
14. Subjects with hereditary disorders including galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption, etc.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of heartburn-free days for 4 weeks (daytime/nighttime) | 4 Weeks

SECONDARY OUTCOMES:
Percentage of major symptom-free (heartburn, acid regurgitation, or heartburn/acid regurgitation) days for 2 and 4 weeks (daytime/nighttime, daytime and nighttime) | 4 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Wonkwang University Hospital, Iksan, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No